CLINICAL TRIAL: NCT03809481
Title: Open-Label, Randomised, Active Controlled, Multi-Centre Ph 3 Study to Evaluate the Safety and Efficacy of Danaparoid vs Argatroban in Acute HIT
Brief Title: Open-Label, Randomised, Active Controlled, Multi-Centre Phase 3 Study Safety and Efficacy of Danaparoid vs Argatroban
Acronym: HITSOVA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Prolonged delay as a result of impact of Covid19 pandemic
Sponsor: Aspen Global Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERGCR-18-ORGHIT-001
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Heparin-induced Thrombocytopenia
MeSH Terms: interventions — danaparoid; argatroban

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, active-controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Danaparoid Sodium (Experimental): Subjects will receive danaparoid via IV infusion for at least 7 days then transition to a VKA. IV loading bolus injection of 2250 U, followed by 400 U/h for 4 hours, then 300 U/h for 4 hours, then a maintenance infusion of 150-200 U/h.
  Interventions: Drug: Danaparoid Sodium
- Argatroban (Active Comparator): Subjects will receive argatroban 2 microgram/kg/min as a continuous infusion, titrated to an aPTT that is 1.5 to 3.0 x initial baseline value, but not exceeding 100 seconds.
  Interventions: Drug: Argatroban

INTERVENTIONS:
Drug: Danaparoid Sodium — inhibits thrombin generation by indirect anti-Xa inhibition and direct inhibition of factor IX activation
  Other Names: Orgaran
  Arms: Danaparoid Sodium
Drug: Argatroban — Synthetic direct thrombin inhibitor
  Arms: Argatroban

SUMMARY:
An Open-Label, Randomised, Active Controlled, Multi-Centre Phase 3 Study to Evaluate the Safety and Efficacy of Danaparoid vs Argatroban in Treatment of Subjects with Acute HIT (HITSOVA study)

DETAILED DESCRIPTION:
Objectives:

Primary:

To show that for the treatment of subjects with acute heparin-induced thrombocytopenia (HIT) danaparoid use is not inferior to argatroban in terms of efficacy. The primary efficacy endpoint (composite endpoint) is defined as treatment response at Day 44.

A subject will be considered a treatment responder, if none of the following events occur by Day 44:

* New or extended venous and/or arterial thrombosis, including gangrene/skin necrosis Note: 'thrombosis' denotes venous and/or arterial here and throughout the protocol
* All-cause mortality
* Unplanned amputation, including ischemic gut resection

Secondary/Exploratory:

To collect additional efficacy data

* Percentage of subjects with increase in platelet count to values ≥ 100,000/ μL at day 14
* Deaths due to TE or bleeding up until Day 44
* Incidence of fatal or non-fatal major bleeding up until Day 44

Note: As outlined by the Control of Anticoagulation Subcommittee major bleeding in non-surgical subjects is defined as:

1. Fatal bleeding, and/or
2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or
3. Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/ L) or more, or leading to transfusion of two or more units of whole blood or red cells

   * New or extended thrombosis, including gangrene/skin necrosis
   * Unplanned amputation, including ischemic gut resection
   * All-cause mortality

Exploratory

* Time to first event (new/extended thrombosis, all cause mortality, unplanned amputation)
* Time to reach consistent increase in 3 consecutive alternate day platelet count measurements during acute treatment
* Incidence of new or extended TE events, including gangrene/skin necrosis up until Day 14
* Incidence of all-cause mortality up until Day 14
* Incidence of unplanned amputation up until Day 14
* Incidence of fatal or non-fatal major bleeding up until Day 14

To describe the safety of danaparoid in comparison to argatroban

* All-cause mortality
* Incidence of fatal and non-fatal major bleeding events (as defined above) during the acute treatment and then the entire follow-up period (until Day 44)
* Incidence of serious adverse events (SAEs)
* Incidence of adverse events (AEs)
* Changes in vital parameters (heart rate, blood pressure, and respiratory rate) and 12-lead electrocardiogram (ECG)
* Incidence of positive pre-danaparoid cross reactivity in the Heparin-induced Platelet Activation (HIPA) assay (Greinacher. 1991)
* Safety laboratory parameters

Design:

This is a Phase 3, open-label, randomized, active-controlled, multi-center study to evaluate the safety and efficacy of danaparoid versus argatroban in treatment of subjects with acuteHIT.

Subjects who develop a reduction in platelet count (PC) greater than or equal to 30% compared with the higher of their pre-heparin treatment count or their highest platelet count after the start of heparin either

1. Between Days 4 and 14 of the start of heparin treatment with or without thrombosis or
2. At Day 1 of heparin treatment and recent heparin exposure (within the last 30 days with or without thrombosis) and who have a score on the 4Ts test of >3 will be considered for study enrollment as a Suspected HIT.

Subjects who have tested negative in available screening tests for HIT within the last 48 hours before enrollment will not be considered for study enrollment, unless new clinical symptoms occurred.The following will occur for all subjects (regardless of whether they had a screening HIT test performed in the enrolling hospital or not):

1. All heparin administration must be ceased after strong clinical suspicion of HIT, based on clinical evaluation of the subject, including the use of heparin-bonded vascular access catheters and circuits as well as heparin flushes.
2. Subject must be randomized into the study and treated with the study drug or transferred to alternative non-heparin anticoagulant in situations where study drug cannot be started within 2 hours after stop of heparin.
3. A blood sample may be taken at the same time for HIT testing according to local practice.
4. The investigator will assess the subject for eligibility for the HITSOVA study by clinical criteria (4T score >3) and inclusion and exclusion criteria.
5. If eligible, written informed consent will be obtained from the subject or a legal guardian and the subject will be randomized to receive study drug. .
6. A new blood sample for HIPA/ PF4/heparin IgG ELISA and anti-danaparoid antibodies and cross reactivity has to be obtained to allow consistent blood sample labelling and documentation before start of study drug, regardless whether another blood sample for HIT testing according to local practice had been obtained at the time of suspicion of HIT

Note, although use of non-heparin treatment for suspected HIT is allowed before enrollment of the subject into the HITSOVA study, the study drug should be started as soon as possible, but no later than 48 hours. In such situation, all time points specified in this protocol, will be calculated from the time of first dose of study drug.

HIT diagnosis will be confirmed serologically by the HIPA assay and a specific PF4/heparin IgG ELISA test for the HIT IgG by the nominated central laboratory based in Greifswald, Germany Subjects with a positive HIPA assay and a positive HIT IgG antigen test with optical density (OD) > 0.5 will be classified as confirmed HIT, and treatment with randomized study drug will continue.Subjects with negative HIPA assay and a positive HIT IgG antigen test with an optical density (OD) >0.5 and subjects with a positive HIPA assay but a negative HIT IgG antigen test OD ≤0.5 will be classified as suspected HIT and treatment with randomized study drug will continue. These subjects will later be adjudicated retrospectively by the Adjudication Committee (AdjC) and then grouped into highly likely HIT or non-HIT.

All other subjects will be considered as non-HIT and the subjects will be removed from the protocol, study drug will be discontinued, and further procedures and treatment will be given at the discretion of the Investigator according to local standard practice. These subjects will be followed to Day 44 after their first dose of study drug for assessment of safety.

During the treatment period if it becomes necessary for an operation, invasive vascular procedure or acute kidney injury requiring the use of an extracorporeal circulation machine develops, then specific dosing instructions are available.

If the acute kidney injury does not recover during the treatment period and the use of an extracorporeal circulation machine is required longer, then the subject will not be eligible to be included in the per protocol set (PPS), but will still be eligible to be included in the full analysis set (FAS).

Study Population:

All subjects who develop a reduction in platelet count (PC) ≥ 30% compared to the higher of their pre-heparin treatment count or their highest platelet count after the start of heparin at either

a) between Days 4 and 14 of the start of heparin treatment with or without thrombosis or b) at Day 1 of heparin treatment (and recent heparin exposure within the last 30 days) with or without thrombosis and who have a score on the 4Ts test of >3 and who are later suspected HIT by the HIPA assay or HIT IgG..

Clinical signs of HIT are

* New thrombosis, on either side (arterial or venous) of the circulation
* Acute systemic reaction when heparin infusion was given:

  * Fever
  * Chills
  * High blood pressure
  * Tachycardia
  * Shortness of breath
  * Chest pain
* Transient global amnesia
* White clot syndrome
* Skin necrosis
* Occlusion of an extracorporeal circuit

Pediatric subjects will not be included in every country in this study. The countries that allow inclusion of pediatric patients are France, USA,and Italy.

It is anticipated that some subjects will be dosed with alternative non-heparin anti-coagulants prior to completing enrollment steps for this study. These subjects can be enrolled in the study as long as the exposure to those treatments is less than 48 hours.

Baseline/screening (Day 0) and enrollment into the study (Day1) can occur on the same day. In this case the assesments for Day 0 and Day 1, should only be performed once.

ELIGIBILITY:
At the time of enrollment subjects are eligible to be included in the study only if all of the following criteria apply:

1. Signed written informed consent by the subject who is able to assess the nature, significance and scope of the clinical trial. If the subject is in emergency situation and temporarily incapable of consent, the consent of a legal representative or authorized representative will be waived if permitted under applicable local regulations/ethics committee recommendations. Consent must be obtained for further participation in the clinical trial as soon as this is possible and reasonable for the subject to do so to confirm understanding/willingness to participate in the clinical study and ability to comply with study procedures and the study visit schedule.
2. Males or females aged ≥2 weeks
3. Subjects with suspected HIT by 4Ts of >3 and with reduction of platelet count of ≥ 30% at either:

   1. Between Day 4 and 14 of the start of heparin exposure or
   2. At Day 1 of heparin exposure with pre-treatment with heparin within the last 30 days, with or without thrombosis.
4. Have adequate renal function: estimated glomerular filtration rate (eeGFR) ≥ 15 mL/min/1.73 m²
5. Male participants:

   A male participant must agree to use contraception during the treatment period and for at least 5 days after the last dose of study intervention and refrain from donating sperm during this period.
6. Female participants: female participant is eligible to participate if 1 of the following conditions applies:

Not a woman of childbearing potential or A woman of childbearing potential who agrees to follow the contraceptive guidance during the treatment period and during the entire VKA use and for one month after cessation of its use. Subjects should continue with adequate contraception after the study end if they continue with VKA use. (Subjects taking oral contraceptives or hormone replacement therapy must have a stable dose and regimen for ≥ 3 months prior to entry into the study.)

Exclusion Criteria:

At the time of enrollmentsubjects are excluded from the study if any of the following criteria apply:

1. Premature infants (corrected age <37 weeks gestational age)
2. Subjects undergoing Extracorporeal Membrane Oxygenation (ECMO) treatment
3. Fibrinolytic therapy <24 hours before enrollment
4. Lumbar puncture or spinal/epidural catheter placement within the past 48 hours
5. Severe hepatic impairment (Child-Pugh Class C) Note: in patients with suspected/confirmed severe liver disease, Child-Pugh C stage of liver disease must be excluded before start of treatment. For calculating Child-Pugh score, laboratory parameters in the patient file on INR, prothrombin time, serum albumin and total bilirubin taken can be taken, if they have been obtained within the last 48 hours before randomization. In all other patients these parameters have to be measured before start of treatment to identify potential exclusion criteria.
6. Active bleeding
7. Subjects with the following conditions to be excluded if alternative antithrombotic treatments are available:

   (i) Severe hemorrhagic diathesis, (ii) Traumatic damage to the central nervous system (iii) Brain, spinal or ophthalmologic surgery (iv) Active stomach/duodenal ulcers or active peptic ulcer unless this ulcer is the cause of the surgical procedure
8. An unexplained activated partial thromboplastin time (aPTT) > 2 x the normal range
9. A hemorrhagic cerebrovascular accident within the previous 3 months
10. Severe, uncontrolled hypertension defined as blood pressure >180/110 mmHg
11. Diabetic retinopathy
12. Acute bacterial endocarditis
13. Expectation of a long-term (> 3 weeks) hemodialysis requirement before the end of the acute treatment
14. Hypersensitivity to the active substances or to any of the excipients
15. Hypersensitivity to sulphite
16. Any investigational drug(s) use within 4 weeks preceding screening or anticipated use during the course of the study
17. Pregnant or breastfeeding woman
18. Use of intra-aortic balloon pump, or ventricular assist device
19. Use of any non-heparin anticoagulant treatment for suspected HIT for more than 48 hours before enrollment.

Ages: 2 Weeks to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Composite Efficacy Response | Day 44
  Efficacy will be assessed by the number of subjects with suspected HIT who respond to treatment. A responder is defined as a subject who has not experienced any of the following from Day 1 to Day 44:
  1. New or extended venous and/or arterial thrombosis, including gangrene/skin necrosis
  2. All-cause mortality
  3. Unplanned amputation, including ischemic gut resection
  Efficacy endpoints as defined above will be assessed by clinical exam with special attention to assessments for thromboses, gangrene, and skin necrosis. Clinically suspected thrombosis will be confirmed/ruled out by objective measures, e.g. compression ultrasound.

SECONDARY OUTCOMES:
Consistent increases in platelet count | Days 14
  Percentage of subjects with increase in platelet count to values ≥ 100,000/ μL
Death due to TE or bleeding | Day 44
  Death due to TE or bleeding
Major Bleeding | Day 44
  Incidence of fatal or non-fatal major bleeding
New or extended thrombosis | Day 44
  New of extended thrombosis, including gangrene/skin necrosis
Unplanned amputation | Day 44
  Unplanned amputation, including ischemic gut resection
All-cause mortality | Day 44
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (35):
- United States (5):
  - Shands University of Florida, Gainesville, Florida
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Bosnia and Herzegovina (5):
  - Clinical Center of the Republic of Srpska, Medical Intesnive Care Unit, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska, Clinic for cardiology, Banja Luka
  - University Clinical Centre of the Republic of Srpska, Lung Clinic, Banja Luka
  - Clinical Center University of Sarajevo, Clinic for Heart, Blood Vessels and Rheumatic Diseases, Sarajevo
  - Clinical Center University of Sarajevo, Clinic for Lung Diseases, Sarajevo
- Jewish General Hospital, Montreal, Canada
- France (3):
  - CHU St Etienne; Avenue Albert Raimond, Saint-Priest-en-Jarez, Auvergne-Rhône-Alpes
  - DIJON University Hospital, Dijon, Burgundy
  - Centre Hospitalier Universitaire Amiens Picardie, Amiens, Somme
- Germany (6):
  - Vivantes Klinikum im Friedrichhain Hämophiliezentrum, Gerinnungssprechstunde Landsberger Allee 49, Berlin, Berlin-Brandenburg
  - Universitätsklinikum Gießen und Marburg GmbH, Klinik für Herz-, Kinderherz- und Gefäßchirurgie Standort Gießen, Giesen, Lower Saxony
  - Städtisches Klinkum Dresden, Dresden, Saxony
  - Universitatstklinikum Halle (Saale), Medizinische Klinik III, Halle, Saxony-Anhalt
  - University Hospital Greifswald Dpt. of Hematology, Greifswald
  - Zentrum für Klinische Transfusionsmedizin, Tübingen
- Italy (4):
  - Azienda Ospedaliero Universitaria S.Orsola-Malpighi - UO Angiologia e Malattie della Coagulazione, Bologna, Emilia-Romagna
  - AOU Careggi, SOD Malattie Aterotrombotiche, Florence, Florence
  - ASST Papa Giovanni XIII, Servizio di Immunoematologia e Medicina Trasfusionale, Bergamo, Lombardy
  - Instituto Scientifico San Raffaele- Servizio Coagulazione e Centro Trombosi, Milan
- Poland (2):
  - Centrum Medyczne HCP Sp. z o.o. Szpital im. Św. Jana Pawła II, Poznan
  - Wojewódzki Szpital Zespolony im. L. Rydygiera, Torun
- Russia (5):
  - First City Hospital N.A. E.E. Volosevich, Arkhangelsk
  - Moscow City Hospital 67, Moscow
  - Oncology Center, Omsk
  - Regional Hospital after N.N Burdenko, Penza
  - Clinical Hospital № 122 N. A. L.G. Sokolov, Saint Petersburg
- Serbia (4):
  - The Institute for Pulmonary Disease of Vojvodina, Pulmonary thromboembolism department, Novi Sad, Sremska Kamenica
  - Clinical Centre of Serbia, Clinic for Emergency Internal Medicine, Belgrade
  - Clinical centre of Serbia, Clinic for Pulmonology, Belgrade
  - Instiute of Cardiovascular Diseases "Dedinje", Belgrade

IPD SHARING:
Plan to Share IPD: No